CLINICAL TRIAL: NCT05722847
Title: Development of an Enhanced Risk Stratification System for Patients With Hospital-diagnosed Advanced Lung Cancer
Brief Title: Risk Stratification for Patients With Hospital-diagnosed Advanced Lung Cancer
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2205
Record Dates: First submitted 2023-01-26; First posted 2023-02-10 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer
Keywords: Advanced Cancer; High-Risk; patient reported outcome
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low risk: Subjects will be considered low risk if they have non-small cell histology, a length of hospital stay <= 8 days, no or low comorbidity, no emergency department use or hospitalization in the 6 months prior, no wheelchair requirement when hospital discharge, or other than Black and/or Hispanic race.
- High risk: Subjects will be considered high risk if they have small cell histology, a length of hospital stay > 8 days, high comorbidity, emergency department use or hospitalization in the 6 months prior, prescription of a wheelchair when hospital discharge, or Black and/or Hispanic race.
- Health Care Providers Group: Thoracic medical oncology physicians, advance practice providers, and nurse navigators respond to the survey that assess acceptability.

SUMMARY:
This study explores whether supportive care interventions that might reduce rehospitalization could be implemented and feasible, in subjects within a high-risk group of subjects with newly diagnosed hospitalized advanced lung cancer (ALC).

This study screened 50 subjects from health records and consented to 15 of these screened subjects. These 15 subjects responded to PRO questionnaires.

DETAILED DESCRIPTION:
Subjects will be considered high risk if they have small cell histology, longer than 8 days hospitalization, high comorbidity, emergency department use or hospitalization in the previous 6 months, prescription of a wheelchair on hospital discharge, or Black and/or Hispanic race. Supportive care interventions such as navigation and palliative care will be recommended for this group.

All hospitalized subjects with newly diagnosed ALC will be offered web- or telephone-based patient-reported outcome (PRO) symptom monitoring for 90 days following hospital discharge if they provide consent. Medical record evaluation of consented subjects will provide data for risk assessment and the high-risk group definition. Healthcare utilization including emergency department visits, hospitalizations, outpatient palliative care, and cancer treatment received will be compared.

ELIGIBILITY:
Inclusion Criteria for Patient Participants:

1. Age ≥ 18 years at the time of screening.
2. Hospital-diagnosed Advanced lung cancer with histological confirmation of disease or suspected lung cancer in the opinion of the treating oncologist.

For PROs only

1. Able to complete a web-based or telephonic symptom survey.

Exclusion Criteria for Patient Participants:

1. Enrollment in hospice upon discharge from the index hospitalization For PROs only

1. Inability to read or speak English.
2. Dementia, altered mental status, or any psychiatric condition as determined by the clinical or study team that would prohibit the understanding or rendering of informed consent.
3. Current incarceration.
4. Any condition that would prohibit the patient from completing PROs

Inclusion Criteria for Health Care Provider Participants:

1. Thoracic medical oncology physicians, advance practice providers, and nurse navigators work in the study site and respond to the survey that assesses acceptability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study has 2 different populations: Patient participants and Health Care Providers. Subjects with hospital-diagnosed advanced lung cancer must meet all of the eligibility criteria, and Health Care Workers provide care to these subjects.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Success of the risk-based stratification system implementation - contacted | Up to 5 days
  The success of the risk-based stratification system implementation- contacted will be determined by the ratio of subjects who were contacted to the whole group is equal to or higher than 70%, in the high-risk group.
Success of the risk-based stratification system implementation - referred | Up to 5 days
  The success of the risk-based stratification system implementation- referred will be determined by the ratio of subjects who were referred to the whole group is equal to or higher than 70%, in the high-risk group.
Success of the risk-based stratification system implementation - navigation | Up to 16 days
  The success of the risk-based stratification system implementation- navigation will be determined by the ratio of subjects who received guidance to the whole group is equal to or higher than 70%, in the high-risk group.
Success of the risk-based stratification system implementation - palliative care | Up to 16 days
  The success of the risk-based stratification system implementation - palliative care will be determined by the ratio of subjects who received palliative care to the whole group is equal to or higher than 70%, in the high-risk group.

SECONDARY OUTCOMES:
Time to receipt of outpatient palliative care | Up to 90 days
  The time to receipt of outpatient palliative care will be defined as the time between the date of palliative care and hospital discharge based on the high-risk and low-risk groups.
Acceptability of the supportive care intervention | Up to 180 days
  Acceptability of the supportive care intervention will be assessed by the percentage of subjects who attend supportive care consultations as determined through electronic health records ( EHR) review.
Acceptability of the risk stratification system the time to complete for providers | Up to 90 days
  Acceptability of the risk stratification system time to complete for providers will be assessed by the time to complete risk stratification per subject.
Acceptability of the risk stratification system time to complete thoracic oncology clinical team | Up to 90 days
  Acceptability of the risk stratification system time to complete the thoracic oncology clinical team will be assessed by the perceived usefulness to the thoracic oncology clinical team
Implementation of PRO-based symptom monitoring | Up to 90 days
  Implementation of patient reported outcomes (PRO)-based symptom monitoring will be determined by the percentage of eligible subjects who complete weekly PROs and the percentage of concerning symptoms reported to the clinical team of more than 70.
Implementation of PRO-based symptom monitoring reported to clinical team | Up to 90 days
  Implementation of PRO-based symptom monitoring will be determined by the percentage of concerning symptoms reported to the clinical team.
Acceptability of PRO-based symptom monitoring subject | Up to 90 days
  Acceptability of PRO-based symptom monitoring to subjects will be measured by the percentage of eligible subjects who agree to participate in the patient-reported outcome report (PRO) system (success: >66%).
Acceptability of PRO-based symptom monitoring to the clinical team | Up to 90 days
  Acceptability of PRO-based symptom monitoring to the clinical team will be determined by the percentage of concerning symptoms resulting in action by any member of the clinical team.(success: >75% reporting somewhat useful, useful, or very useful).
Acceptability of PRO-based symptom monitoring to the thoracic oncology clinical team | Up to 90 days
  Acceptability of PRO-based symptom monitoring to the clinical team will be determined by the percentage of concerning symptoms perceived usefulness to the thoracic oncology clinical team (success: >75% reporting somewhat useful, useful, or very useful).

CONTACTS AND LOCATIONS:
Overall Officials: Emily Ray, MD, Principal Investigator — Lineberger Comprehensive Cancer Center, The University of North Carolina Chapel Hill
Locations (1):
- UNC Lineberger, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials